CLINICAL TRIAL: NCT00742183
Title: An Open, Parallel, Randomized, Comparative, Multi-centre Investigation in US Evaluating the Cost-effectiveness, Efficacy, Safety and Tolerance of Mepilex® Ag Versus Silvadene® in the Treatment of Partial Thickness Burns.
Brief Title: Evaluating the Cost-effectiveness, Efficacy, Safety and Tolerance of Mepilex® Ag Versus Silvadene®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PUMA 415
Record Dates: First submitted 2008-08-19; First posted 2008-08-27 (Estimated); Results first posted 2010-11-19 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-11

CONDITIONS: Second Degree Burn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mepilex® Ag (Experimental): Mepilex® Ag consists of a Safetac® soft silicone wound contact layer, a grey absorbent polyurethane foam pad containing a silver compound, activated carbon, and a vapour permeable waterproof film. Mepilex® Ag is an antimicrobial soft silicone foam dressing that absorbs exudate and maintains a moist wound environment.
  Mepilex® Ag contains silver sulphate that releases silver ions to inactivate a wide range of wound related pathogens (bacteria and fungi), shown in vitro. By reducing the number of microorganisms, Mepilex® Ag may also reduce odour.
  Interventions: Device: Mepilex
- Silvadene® Cream 1% (Active Comparator): Silvadene® Cream 1% (silver sulfadiazine) is a topical antimicrobial drug indicated as an adjunct for the prevention and treatment of wound sepsis in patients with second-and third-degree burns.
  Interventions: Device: Silvadene

INTERVENTIONS:
Device: Mepilex — Mepilex Ag - dressing changes every 5-7 days, more frequently if needed
  Arms: Mepilex® Ag
Device: Silvadene — Silvadene - dressing changes every day, more frequently if needed
  Arms: Silvadene® Cream 1%

SUMMARY:
The primary objective is to compare the incremental costs (direct and indirect) and benefits (healing outcomes, quality of life) of using foam silver dressing (Mepilex® Ag) to a Silver sulfadiazine 1% cream (Silvadene®) from the perspective of the health care provider.

The secondary objectives are to investigate the safety, the tolerance and the performance on burn status including pain.

DETAILED DESCRIPTION:
In- and/or out-patients at ten centers in the United States were included in this investigation. Subjects included were 5 years of age and older who suffered from partial thickness burns. Every patient was followed for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a second degree burn covering 5% to 20% BSA. TBSA covered with burn is allowed to be up to 25%, allowing a maximum of 10% to be third degree burn (only the Second degree burn should be treated)
* Burn of thermal origin
* Both gender with an age ≥ 5 years at randomization
* Signed informed consent
* Subjects who are younger than the legal consenting age must have a legally authorized representative

Exclusion Criteria:

* - Burns equal to or older than 36 hours
* Burns of chemical and electrical origin
* Clinically infected Burn (as judged by the investigator)
* Treatment of the burn with an active agent before study entry, SSD is allowed up to 24 hours prior to randomization
* Patients with necrotising leucocytic vasculitis or pyoderma gangrenosa.
* Diagnosed underlying disease(s) (e.g. HIV/AIDS, cancer and severe anaemia) judged by the investigator to be a potential interference in the treatment.
* Patients with insulin dependent diabetes mellitus
* Patients treated with systemic glucocorticosteroids, except patients taking occasional doses or doses less than 10mg prednisolon/day or equivalent.
* Use of immunosuppressive agents, radiation or chemotherapy within the past 30 days.
* Known allergy/hypersensitivity to any of the components of the investigation products.
* Patients with physical and/or mental conditions that are not expected to comply with the investigation.
* Participation in other clinical investigation(s) within 1 month prior to start of the investigation
* Pregnancy
* Previously randomised to this investigation

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-08; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Silverstein, Principal Investigator — Paul Silverstein Burn Center
Locations (10):
- United States (10):
  - LA County Hospital & USC Medical Center, Los Angeles, California
  - The Burn Center, Washington Hospital Center, Washington D.C., District of Columbia
  - Shands Burn Center, University of Florida, Gainesville, Florida
  - Joseph Still Burn Center, Augusta, Georgia
  - UI Burn Treatment center, Iowa City, Iowa
  - Cornell Medical Center, New York, New York
  - Paul Silverstein Burn center, Oklahoma City, Oklahoma
  - St Christopher's Hospital, Philadelphia, Pennsylvania
  - Southwestern Regional Burn Center, Parkland Hospital, Dallas, Texas
  - Department of Surgery, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Investigation period: Sept 2008 - Sept 2009. In- and/or out-patients at ten centers in US were included in this investigation. Subjects included were 5 years and above and suffered from partial thickness burns.
Groups:
- Mepilex Ag: Treatment period will be a maximum of three weeks with Silvadene® or Mepilex® Ag.
  Dressing changes of Mepilex® Ag will be performed every 5-7 day, depending on the status of the burn
- Silvadene: Silver sulfadiazine 1% cream treatment period will be a maximum of three weeks. Dressing changes of Silvadene® will be performed at least once per day.
Period: Overall Study
Arm/Group | Mepilex Ag | Silvadene
Started | 49 (50 subjects randomised, one of them did not receive any treatment.) | 51
Completed | 40 | 39
Not Completed | 9 | 12
Not completed — Adverse Event | 2 | 2
Not completed — Death | 1 | 0
Not completed — Physician Decision | 0 | 2
Not completed — Lost to Follow-up | 4 | 4
Not completed — Required skin-graft | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lack of Efficacy | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Mepilex® Ag: The dressing to be used Mepilex® Ag, consists of an absorbent polyurethane foam pad containing silver sulphate with a silicone contact layer with the Safetac® technology. The silver ions are hydro activated in presence of fluid or wound exudates.
- Silvadene® Cream 1%: Silvadene® Cream 1%, silver sulfadiazine is a topical antimicrobial drug indicated as an adjunct for the prevention and treatment of wound sepsis in patients with second-and third-degree burns.
- Total: Total of all reporting groups
Arm/Group | Mepilex® Ag | Silvadene® Cream 1% | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 4 | 8
  Between 18 and 65 years | 41 | 41 | 82
  >=65 years | 4 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (18.1) | 39.2 (18.2) | 38.4 (18.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 36 | 41 | 77
Region of Enrollment [Number; unit: participants]
  United States | 49 | 51 | 100

OUTCOME MEASURES:

1. Primary Outcome: Compare the Costs of Using the Interventions (Direct and Indirect)
Description: The incremental cost-effectiveness ratio is calculated as the difference in total costs in each group divided by the difference in rate of full re-epithelialization (taken from the survival curve) at 20 days in each group (Δcosts/ Δeffects). Total costs were calculated based on the costs of primary and secondary dressings, silver sulphadiazine cream and estimated application, labor, supplies and pain medications. These costs were estimated from a representative sample of each population, across study facilities, using activity-based costing methods.
  The incremental cost-effectiveness ratio is interpreted as the price of additional health benefits. The ratio is supposed to be used by decision makers, in order for them to compare their willingness-to-pay for an additional health benefit with the pr
Time Frame: August 2008-August 2009
Population: Primary analysis: the Intention To Treat (ITT) population will include all patients subject to at least one post-randomisation treatment and that provide some data for the primary endpoint. If there are any patients included which do not comply with the inclusion/exclusion criteria they will be included in the ITT population
Measure: Mean (95% Confidence Interval); unit: dollars
Groups:
- Mepilex Ag; Silvadene: Patients with a second degree burn covering 5% to 20% BSA. TBSA covered with burn is allowed to be up to 25%, allowing a maximum of 10% to be third degree burn (only the Second degree burn should be treated).
Arm/Group | Mepilex Ag | Silvadene
Number analyzed (Participants) | 49 | 51
dollars | 395.03 [343.68 to 450.30] | 775.79 [659.42 to 892.16]

ADVERSE EVENTS:
Groups:
- Mepilex Ag: Mepilex® Ag is an antimicrobial soft silicone foam dressing that absorbs exudate and maintains a moist wound environment.
- Silvadene: Silvadene® Cream 1%, silver sulfadiazine is a topical antimicrobial drug.
Arm/Group | Mepilex Ag | Silvadene
Serious Adverse Events (participants affected / at risk) | 2/49 | 1/51
Other Adverse Events (participants affected / at risk) | 20/49 | 26/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepilex Ag (N=49) | Silvadene (N=51)
Death (General disorders) | 1 (1) | 0 (0) — Patient died, description of SAE was Acute Bronco spasm. The patient had a history of CHF. Relationship to investigation product judged as unlikely
Pain (General disorders) | 0 (0) | 1 (1)
Anticoagulation drug level above therapeutic (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepilex Ag (N=49) | Silvadene (N=51)
Constipation (Gastrointestinal disorders) | 5 (5) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 4 (4)
Nausea (Gastrointestinal disorders) | 8 (8) | 10 (10)
Staphylococcal infection (Infections and infestations) | 4 (4) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 12 (12)
Skin graft (Surgical and medical procedures) | 2 (2) | 4 (4)
Hypertension (Vascular disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Coordinating Investigator will be the lead author for the mail (primary) publication from this Investigation. For any abstract and/or manuscript the Investigators will be given at least 14 days review time before the intended submission of the document.